CLINICAL TRIAL: NCT05067400
Title: SARS-CoV-2 (COVID-19) Antibody PrevalencE in an Adult London HIV Cohort
Acronym: SCAPE-HIV
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-09-29; First posted 2021-10-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: HIV-1-infection; SARS-CoV Infection; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational SARS-CoV2 serological surveillance single London HIV outpatient center study using NHS participants

DETAILED DESCRIPTION:
The main aim of this study is to find out how many people living with HIV (PLWH) attending a major HIV centre in London, have already been infected with SARS-CoV2 so far which will be determined through serological blood tests detecting the presence of antibodies to SARS-CoV2, or have developed antibodies in response to vaccination.

However, it is not know whether the presence of antibodies from natural infection means anything more than a marker that someone has been exposed to SARS-CoV2 previously. It is not know whether this means someone is any less likely to be reinfected in the future or how it will affect possible future infections with SARS-CoV2. Whilst further data on natural and vaccine induced antibody responses is awaited, those with the presence of anti-SARS-CoV2 antibodies continue to be advised to take the same precautions as everyone else in terms of reducing the risk of getting COVID-19: regularly washing hands, wearing a mask and remaining socially distant where possible.

Now that vaccination has commenced it is also unclear what markers of vaccine induced immunity will develop, including in PLWH. This study will help better determine whether HIV should be an additional 'priority' group for vaccination, and also what antibody responses exist in PLWH who have been vaccinated

The intention is to invite the cohort in for an annual set of HIV related blood tests, covering those who are scheduled for bloods, as well as those who may have missed scheduled blood monitoring appointments during the COV19 lockdown period. In addition to these tests the study proposes offering serological testing for SARS CoV-2 as part of this surveillance study. Participation will be voluntary, and informed consent will be obtained. Participants will be informed of their result along with information about the uncertainty of its meaning, beyond indicating previous infection or vaccination.

The study aims to test for the presence of specific antibodies that target SARS-CoV2 in people living with HIV, as a marker of whether someone has been infected before. This will help create a better understanding of whether living with HIV puts people at a higher risk of becoming infected with SARS-CoV2 compared to the general population, and which other factors or characteristics may affect this risk. This will help identify who might be more at risk of getting COVID-19 in the future and will help plan for future COVID-19 vaccine strategies.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Registered patient at ICDC
* Age ≥18 years at study entry
* Able to comprehend study patient information leaflet

Exclusion Criteria:

* Unable to give informed consent and participant without a good understanding of verbal and written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive participants attending the Ian Charleson Day Centre clinic (ICDC) at the Royal Free Hospital, London for their HIV care.
  Population aged 18+ years
Sampling Method: Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV2 antibodies | Since 1st Jan 2020
  The primary outcome measure is the presence of antibodies to SARS-CoV2. This is a binary outcome (present/absent)

SECONDARY OUTCOMES:
Reporting of COVID symptoms | Since 1st Jan 2020
  The secondary outcome measure is the reporting of previous COVID symptoms since 1st January 2020. This is a binary measure (yes/no).

OTHER OUTCOMES:
Reporting of previous SARS-CoV2 infection (reported history) | Since 1st Jan 2020
  Reported history of positive SARS CoV2 test since 1 Jan 2020
History of SARS CoV2 vaccine | Since 1st Jan 2020
  Reported history of receiving a SARS CoV2 vaccine (no, 1 dose, 2 dose)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Barber, MBBChir, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No